CLINICAL TRIAL: NCT03388268
Title: Double Blinded, Randomized Controlled Trial of Oral Vancomycin Versus Placebo in Hospitalized Patients With Diarrhea and Stool toXin NEGative But Nucleic Acid Amplification Test Positive for Toxigenic Clostridium Difficile (TOX NEG Trial)
Brief Title: TOX NEG Trial: Clostridium Difficile Diagnosis and Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 201708055
Record Dates: First submitted 2017-12-05; First posted 2018-01-02 (Actual); Results first posted 2021-07-23 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Clostridium Difficile Infection; Diarrhea
Keywords: Clostridium difficile; Diarrhea
MeSH Terms: conditions — Clostridium Infections; Diarrhea | interventions — Vancomycin

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized controlled trial of CDI treatment with oral vancomycin vs. placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Oral vancomycin (Active Comparator): 125mg of oral vancomycin four times per day
  Interventions: Drug: Oral Vancomycin; Device: Toxin enzyme immunoassay; Device: Nuceleic acid amplification test
- Placebo (Placebo Comparator): Placebo four times per day
  Interventions: Drug: Placebo; Device: Toxin enzyme immunoassay; Device: Nuceleic acid amplification test

INTERVENTIONS:
Drug: Oral Vancomycin — Oral vancomycin 125mg 4 times per day
  Other Names: Vancocin
  Arms: Oral vancomycin
Drug: Placebo — Sugar liquid manufactured to mimic oral vancomycin 125mg
  Arms: Placebo
Device: Toxin enzyme immunoassay — EIA assay: Wampole/Tech Lab Tox A/B II
Device: Nuceleic acid amplification test — NAAT: Xpert C. difficile, Cepheid

SUMMARY:
The purpose of this study is to determine the risks and benefits of antibiotic treatment for Clostridium difficile infection (CDI) among patients whose stool samples are nucleic acid amplification test (NAAT) positive and enzyme immunoassay (EIA) negative for C. difficile.

Currently, healthcare facilities use a wide variety of tests and strategies for identifying patients with CDI; both EIA and NAAT are widely used. There is no clear gold standard for identifying CDI. At WUSM and BJH, patients are only treated for CDI if they have a positive EIA. However, at many other healthcare facilities, the standard of care is to treat for CDI if the patient is NAAT positive. Some patients who are NAAT-positive may not have true CDI; while this treatment is standard of care at many facilities, the risk and benefits of treating these patients for CDI is unknown.

We propose to perform a double blinded, randomized controlled non-inferiority trial of antimicrobial of patients who are EIA negative, NAAT positive to determine the risks and benefits of CDI treatment in this population.

DETAILED DESCRIPTION:
Study Purpose:

The purpose of this study is to determine the risks and benefits of antibiotic treatment for Clostridium difficile infection (CDI) among patients whose stool samples are nucleic acid amplification test (NAAT) positive and enzyme immunoassay (EIA) negative for C. difficile.

Background:

Clostridium difficile infection (CDI) is the most common cause of healthcare-associated diarrhea. There is no gold standard diagnostic test for (CDI). Commercially available assays detect C. difficile or its toxins in stool. Nucleic acid amplification tests (NAAT) are much more sensitive than toxin enzyme immunoassays (EIA). However, clinical correlation is needed to determine who has CDI. Most US clinical microbiology laboratories have adopted NAATs for C. difficile under the presumption the enhanced analytical sensitivity was beneficial. Although some patients with NAAT-positive/toxin-negative stool have CDI and a false-negative toxin EIA, subsequent studies indicate most patients with NAAT-positive / toxin-negative stool do not have CDI. Rather, they are asymptomatic C. difficile carriers who have diarrhea for other reasons. Most of these studies also have limitations and considerable controversy remains for whether NAATs or toxin EIAs should be used when CDI is suspected.

Treatment of asymptomatic C. difficile carriers is not beneficial, and may result in harm. At hospitals that utilize NAATs, most patients with NAAT-positive / toxin-negative stool receive treatment for CDI. The most common treatments for CDI, metronidazole and oral vancomycin, are highly disruptive of the intestinal microbiome. These antimicrobials create selective pressures that promote the acquisition and proliferation of antimicrobial resistance and multidrug resistant organisms (MDRO), including public health threats such as MDRO Enterobacteriaceae like carbapenem-resistant Enterobacteriaceae (CRE) and extended-spectrum beta-lactamase (ESBL) producing organisms, vancomycin-resistant Enterococcus (VRE), and the latest emerging threat Candida auris. This leads to MDRO infections and MDRO spread to others. Paradoxically, unnecessary treatment for CDI may increase risk for CDI once treatment is stopped contributing to CDI-related adverse events and C. difficile spread to others. Unnecessary CDI treatment potentially harms both that patient and other people. Whether the benefit of treating patients with NAAT-positive/toxin-negative stool that are missed cases of CDI outweighs the risk of treating patients with NAAT-positive/toxin-negative stool that are asymptomatic C. difficile carriers remains unknown.

This study is a double-blinded randomized controlled trial of CDI treatment for patients with NAAT-positive / toxin-negative stool. Such a trial is necessary to understand the risk-benefit of treating these patients for CDI. Patients with NAAT-positive / toxin-negative stool who consent to participate will be randomized to 10 days of oral vancomycin or placebo. Stool and environmental specimens will be obtained at regular time points and interrogated with culturomic and metagenomic methods. Patients will be followed until eight weeks after discontinuation of study drug. These data and specimens will be used to determine the impact of oral vancomycin versus placebo on the microbiome, C. difficile and MDRO colonization, environmental contamination, duration of diarrhea, CDI-related adverse events, and death.

Specific aims and hypotheses:

Specific Aim 1: Determine if there are differences in microbiome disruption and acquisition / persistence of C. difficile and other MDRO carriage in stool among patients with NAAT-positive / toxin-negative stool who are randomized to a 10-day course of oral vancomycin versus placebo.

Hypotheses: Study participants who receive oral vancomycin will have greater disruption of the taxonomic and functional metabolic profiles of the fecal microbiome, increases in antimicrobial resistance genes, acquire more MDRO, and will have greater persistence and abundance of MDRO in stool compared to participants who receive placebo. Participants who receive oral vancomycin will not have detectable C. difficile in stool after completion of study drug, but will be more likely to have C. difficile in stool at week 8 after completion of study drug compared to participants who receive placebo.

Specific Aim 2: Determine if there are differences in C. difficile and other MDRO environmental contamination between treatment groups.

Hypothesis: Study participants who receive oral vancomycin will have less environmental C. difficile contamination but more MDRO contamination compared to participants who receive placebo while receiving study drug. After study drug is completed, those who receive oral vancomycin will have more environmental contamination due to both C. difficile and other MDROs.

Specific Aim 3: Determine if there are differences in CDI-related outcomes between groups.

Hypothesis: There will be no difference in time to resolution of diarrhea or CDI-related outcomes between treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Stool submitted to the BJH microbiology laboratory for C. difficile testing that tests negative for C. difficile toxins (C. difficile Tox A/B II, Alere, Waltham, MA) as part of routine clinical care and positive by NAAT (Xpert C. difficile, Cepheid, Sunnyvale, CA)
* Clinically significant diarrhea (≥3 diarrheal bowel movements per day or ≥1 diarrheal bowel movement plus abdominal pain)
* ≥18 years of age.

Exclusion Criteria:

* The presence of a condition associated with persistent / prolonged / recurrent diarrhea, including, but not limited to:
* Upcoming chemotherapy
* Previous or upcoming bone marrow/hematopoietic stem cell transplant,
* Leukemia: new, not in remission, or receiving chemotherapy
* Inflammatory bowel disease
* Crohn's disease
* Ulcerative colitis
* Microscopic colitis
* Previous total colectomy
* Previous partial colectomy without return to formed bowel movement or previous resection of colon
* Colostomy or ileostomy
* Unable to follow study procedures
* Not expected to survive until study follow-up is complete
* Allergy or intolerance to oral vancomycin
* A history of CDI in the past 3 months
* Alternate infectious etiology for diarrhea
* Receipt of CDI antibiotic treatment (excluding empiric treatment given while pending EIA results)
* Does not provide consent will exclude a patient from participating in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Dubberke, MD, MSPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Derived] Fishbein SRS, Hink T, Reske KA, Cass C, Struttmann E, Iqbal ZH, Seiler S, Kwon JH, Burnham CA, Dantas G, Dubberke ER. Randomized Controlled Trial of Oral Vancomycin Treatment in Clostridioides difficile-Colonized Patients. mSphere. 2021 Jan 13;6(1):e00936-20. doi: 10.1128/mSphere.00936-20. PMID 33441409

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Vancomycin | Placebo
Started | 8 | 7
Completed | 7 | 4
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Vancomycin | Placebo | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Median (Full Range); unit: years] | 66 [37 to 81] | 64 [48 to 77] | 65 [37 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 4 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-white race | 1 | 1 | 2
  White race | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15
Receiving antibiotics at enrollment [Count of Participants; unit: Participants] | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Detectable C. Difficile
Description: Stool specimens will be examined via culture and metagenomic analyses for the presence of detectable C. difficile. Presence will be defined as presence of culturable C. difficile in stool any time after collection of enrollment stool samples.
Time Frame: Through 8 weeks after completion of study drug
Population: 12 of 15 enrolled patients had follow up stool specimens available for analysis. C. difficile was detected in 9 of these 12 during the follow up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Vancomycin | Placebo
Number analyzed (Participants) | 7 | 5
Participants | 5 | 4

2. Secondary Outcome: Number of Participants With Detectable Environmental Contamination
Description: Swabs from participants' home and hospital environments will be examined via culture and metagenomic analyses for the presence and/or persistence of C. difficile and other multidrug resistant organisms.
Time Frame: Through 8 weeks after completion of study drug
Population: 12 of 15 enrolled patients had follow up environmental swabs available for analysis. C. difficile was detected in 9 of these 12 during the follow up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Vancomycin | Placebo
Number analyzed (Participants) | 7 | 5
Participants | 5 | 4

3. Secondary Outcome: Duration of Diarrhea in Study Participants as Defined by Daily Symptoms and Questionnaire Using the Bristol Stool Chart
Description: Duration of diarrhea will be compared between groups. Duration of diarrhea will be assessed daily during study drug using a questionnaire and the Bristol Stool Chart. The Bristol Stool Chart measures stool consistency. Diarrhea will be defined as Bristol Stool Chart types 5-7.
Time Frame: Through 8 weeks after completion of study drug
Measure: Median (Full Range); unit: Days
Arm/Group | Oral Vancomycin | Placebo
Number analyzed (Participants) | 8 | 7
Days | 2 [2 to 13] | 4 [3 to 11]

4. Secondary Outcome: Presence of Other Multidrug Resistant Organisms in the Gut Microbiome of Study Participants
Description: Stool specimens will be examined via culture and metagenomic analyses for the presence of multidrug resistant organisms before and after study drug.
Time Frame: Through 8 weeks after completion of the study drug
Population: 12 of 15 enrolled patients had follow up stool specimens available for analysis. Multidrug organisms were detected in 10 of these 12 during the follow up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Vancomycin | Placebo
Number analyzed (Participants) | 7 | 5
Participants | 6 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected through 8 weeks after completion of the study drug.
Arm/Group | Oral Vancomycin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/8 | 0/7
Other Adverse Events (participants affected / at risk) | 3/8 | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Vancomycin (N=8) | Placebo (N=7)
Volume overload (Endocrine disorders) | 1 (1) | 0 (0)
Hypoxemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Vancomycin (N=8) | Placebo (N=7)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Headache, vertigo, nausea/vomiting (General disorders) | 0 (0) | 1 (1)
Syncope, altered mental status (General disorders) | 1 (1) | 0 (0)
C. difficile EIA positive stool sample (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT03388268/Prot_000.pdf